CLINICAL TRIAL: NCT01599637
Title: A Phase II, Multi-centre, Randomized, Double Blind, Placebo-controlled Study to Determine the Mode of Action of Omalizumab in Patients With Chronic Idiopathic Urticaria (CIU) Who Remain Symptomatic With Antihistamine Treatment (H1)
Brief Title: Mode of Action Study of Omalizumab in Patients With Chronic Idiopathic Urticaria (CIU) Who Fail to Respond to Antihistamine Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CIGE025E2201; 2011-004216-31 (EudraCT Number)
Record Dates: First submitted 2012-01-25; First posted 2012-05-16 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Idiopathic Urticaria
Keywords: Chronic idiopathic urticaria; CIU; Xolair; IGE025; FcεRI; IgE
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- IGE025 (Experimental): Patients will receive omalizumab administered subcutaneously every 4 weeks at the study center.
  Interventions: Drug: IGE025
- Placebo to IGE025 (Placebo Comparator): Placebo administered subcutaneously every 4 weeks at the study center.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IGE025 — Study medication will be supplied as a lyophilized, sterile powder in a single-use, 5-mL vial.
  Arms: IGE025
Drug: placebo — Study medication will be supplied as a lyophilized, sterile powder in a single-use, 5-mL vial.
  Arms: Placebo to IGE025

SUMMARY:
The study is designed to explore the mode of action for omalizumab therapy in patients with chronic idiopathic urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic spontaneous urticaria refractory to H1 antihistamines at Baseline

Exclusion Criteria:

* Clearly defined underlying etiology for chronic urticarias other than CIU (main manifestation being physical urticaria). This includes the following urticarias: Acute, solar, cholinergic, heat, cold, aquagenic, delayed pressure or contact, as well as the following diseases as these diseases may have symptoms of urticaria or angioedema: Urticarial vasculitis, urticaria pigmentosa, erythema multiforme, mastocytosis, hereditary or acquired angioedema, lymphoma, leukemia, or generalized cancer.
* Previous treatment with omalizumab.
* A history or presence of atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus or other skin disease associated with itch.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Germany (4):
  - Novartis Investigative Site, Dresden, Germany
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Münster

REFERENCES:
- [Derived] Metz M, Torene R, Kaiser S, Beste MT, Staubach P, Bauer A, Brehler R, Gericke J, Letzkus M, Hartmann N, Erpenbeck VJ, Maurer M. Omalizumab normalizes the gene expression signature of lesional skin in patients with chronic spontaneous urticaria: A randomized, double-blind, placebo-controlled study. Allergy. 2019 Jan;74(1):141-151. doi: 10.1111/all.13547. Epub 2018 Oct 15. PMID 29974963

RESULTS

PARTICIPANT FLOW:
Groups:
- IGE025: IGE025 administered subcutaneously every 4 weeks at the study center
- Healthy Volunteers: Healthy volunteer data was collected at baseline only. These healthy volunteers did not receive any test treatment. The data collected from these individuals was used to provide a reference to help characterize the levels of skin biopsy markers and were used in the descriptive analyses but not formally compared with the corresponding levels in the treated subjects
Period: Overall Study
Arm/Group | IGE025 | Placebo to IGE025 | Healthy Volunteers
Started | 20 (" started" indicates randomized safety, pharmacodynamics and pharmocokinetics set) | 10 | 10
Completed | 19 | 8 | 10
Not Completed | 1 | 2 | 0
Not completed — administrative problems | 0 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IGE025 | Placebo to IGE025 | Healthy Volunteers | Total
Number analyzed (Participants) | 20 | 10 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (11.02) | 41.1 (7.96) | 36.4 (9.74) | 38.7 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 8 | 10 | 36
  Male | 2 | 2 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 10 | 10 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Observed Values and Absolute Change From Baseline in FceRI Positive Skin Cells: Dermis, Lesional and Non Lesional Skin
Description: Observed values and absolute change in FcεRI positive skin cells: dermis non-lesional and lesional. The primary variable for this study was the relative change from baseline in the high affinity IgE receptor (FcεRI) positive skin cells, based on skin biopsies collected from patients with CIU after 12 weeks of treatment.The values are average of cell numbers derived from counting 5 consecutive microscopic fields. Area counted is 5x 0.196 mm2
Time Frame: Baseline through Day 85 post-treatment
Population: All subjects who received at least one dose of study drug and had evaluable pharmacodynamic (PD) data were included in the PD data analysis. Patients with both baseline and week 12 data were included in this analysis
Measure: Mean (Standard Deviation); unit: FcεRI positive skin cells
Groups:
- Placebo IGE025: Placebo IGE025 administered subcutaneously every 4 weeks at the study center
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
FcεRI positive skin cells
  FcεRI +ve skin cells: dermis lesional D1 (n=19,8) | 18.14 (7.08) | 15.17 (3.11)
  FcεRI +ve skin cells: dermis lesional d85 (n=10,7) | 13.40 (5.88) | 20.19 (8.76)
  FcεRI +ve skin cells:dermis lesional Chge(n=10,6) | -5.42 (7.42) | 3.69 (10.58)
  FcεRI +ve skincells:dermis nonlesional D1(n=19,10) | 18.91 (9.42) | 20.48 (5.54)
  FcεRI +ve skincells:dermis nonlesional D85(n=18,8) | 14.72 (7.56) | 20.81 (7.30)
  FcεRI +ve skincells:dermis nonlesional Chg(n=17,8) | -5.40 (9.06) | -0.07 (9.33)

2. Primary Outcome: Observed Values and Absolute Change From Baseline in IgE Positive Skin Cells: Dermis, Lesional and Non Lesional Skin
Description: Observed values and absolute change in IgE positive skin cells: dermis non-lesional and lesional The primary variable for this study was the relative change from baseline in IgE positive skin cells, based on skin biopsies collected from patients with CIU after 12 weeks of treatment. The values are average of cell numbers derived from counting 5 consecutive microscopic fields. Area counted is 5x 0.196 mm2
Time Frame: Baseline through Day 85 post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IgE positive skin cells
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
IgE positive skin cells
  IgE positive cells, lesional D1 (n=19,8) | 12.93 (8.61) | 15.23 (15.71)
  IgE positive cells, lesional D85 (n=10,7) | 6.73 (7.90) | 12.47 (6.54)
  IgE positive cells, lesional chg(n=10.6) | -5.69 (10.96) | -3.95 (20.76)
  IgE positive cells,non-lesional D1 (n=19,10) | 13.82 (10.21) | 16.59 (9.35)
  IgE positive cells,non-lesional D85 (n=18,8) | 9.80 (11.66) | 18.30 (7.51)
  IgE positive cells,non-lesional Chng (n=17,8) | -4.87 (9.83) | -0.84 (6.18)

3. Secondary Outcome: Correlation of Change From Baseline in IgE Receptor FceRI With Change From Baseline in UAS7 at Week 12 by Treatment, Skin Layer and Lesion Status
Description: Correlation of primary endpoint with The UAS7 which is a composite eDiary-recorded score with numeric severity intensity ratings on a scale of 0-3 (0 = none to 3 = intense/severe) for 1) the number of wheals (hives); and 2) the intensity of the itch. The daily UAS is the average of the morning and evening scores and the UAS7 is the sum of the daily UAS scores over 7 days.UAS7 score: The sum of the daily UAS scores over 7 days. Range: 0-42. If fewer than 7 but at least 4 daily values were non-missing, the remaining values were imputed to be the average. This is equivalent to multiplying the average of the non missing values by 7. UAS7 score: The sum of the daily UAS scores over 7 days. Range: 0-42. A higher score indicates worse disease.
Time Frame: Baseline through Day 85
Population: Efficacy analysis set: Includes all randomized patients who received at least one dose of study drug and have post-randomization efficacy data.
Measure: Number; unit: correlation coefficient
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
correlation coefficient
  Dermis, lesional | 0.3305 | -0.1889
  Dermis, non-lesional | 0.2785 | 0.5057
  Epidermis, lesional | 0.0021 | 0.0101
  Epidermis, non-lesional | 0.0644 | 0.1563

4. Secondary Outcome: Correlation of Change From Baseline in IgE on Positive Skin Cells With Change From Baseline in UAS7 at Week 12 by Treatment, Skin Layer and Lesion Status
Description: as for outcome 3
Time Frame: Baseline through Day 85
Population: as for outcome 3
Measure: Number; unit: correlation coefficient
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
correlation coefficient
  Dermis, lesional | 0.4841 | -0.0952
  Dermis, non-lesional | 0.2759 | 0.4947
  Epidermis, lesional | 0.2190 | -0.1142
  Epidermis, non-lesional | 0.1574 | -0.2310

5. Secondary Outcome: Observed Values and Absolute Change From Baseline in Skin Cell Subsets (CD3, CD4, CD8, Eosinophils, DCs, and Mast Cells) by Parameter, Skin Layer, Lesion Status, Treatment and Visit
Description: The average number of cells derived from counting 5 consecutive microscopic fields. Area counted is 5x 0.196 mm2
Time Frame: Baseline to Day 85
Population: All subjects who received at least one dose of study drug and had evaluable pharmacodynamic (PD) data were included in the PD data analysis. Day 29 was an optional sampling time point in this paramter. The values are average of cell numbers derived from counting 5 consecutive microscopic fields. Area counted is 5x 0.196 mm2
Measure: Mean (Standard Deviation); unit: # positive cells
Groups:
- IGE025; Placebo IGE025: Dosed every 4 weeks up to 12 weeks
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
# positive cells
  CD11c Epidermis Non lesional Baseline (n= 19,10) | 1.06 (1.077) | 1.25 (0.584)
  CD11c Epidermis Non lesional Day 8 (n=19,10) | 1.41 (1.313) | 0.95 (0.920)
  CD11c Epidermis Non lesional D 8(n=18,10) Chge | 0.39 (1.351) | -0.30 (1.255)
  CD11c Epidermis Non lesional D 29(n=4,0) | 1.00 (0.000) | NA (NA) — no observations made
  CD11c Epidermis Non lesional D 29(n=4,0) Chg | 0.70 (0.383) | NA (NA) — no observations made
  CD11c Epidermis Non lesional D 85(n=18,8) | 1.19 (0.806) | 0.53 (0.544)
  CD11c Epidermis Non lesional D 85(n=17,8) Chge | 0.04 (1.216) | -0.84 (0.524)
  CD11c Epidermis Non lesional D 140(n=17,7) | 1.25 (1.630) | 0.58 (0.942)
  CD11c Epidermis Non lesional D 140(n=17,7) Chge | 0.04 (1.216) | -0.75 (0.939)
  CD11c Epidermis lesional baseline (n=19,8) | 1.17 (1.363) | 3.79 (8.028)
  CD11c Epidermis lesional D8 (n=11,10) | 1.63 (1.425) | 1.19 (1.329)
  CD11c Epidermis lesional D8 (n=11,8) Change | 0.39 (1.153) | -2.74 (8.466)
  CD11c Epidermis lesional D29 (n=5,0) | 1.56 (1.609) | NA (NA) — no observations made
  CD11c Epidermis lesional D29 (n=5,0) Change | 0.88 (1.677) | NA (NA) — no observations made
  CD11c Epidermis lesional D85 (n=10,7) | 1.18 (0.577) | 0.46 (0.378)
  CD11c Epidermis lesional D85 (n=10,6) Change | -0.06 (1.234) | -4.06 (9.384)
  CD11c Epidermis lesional D140 (n=6,5) | 0.53 (0.555) | 0.18 (0.171)
  CD11c Epidermis lesional D140 (n=6,5) Change | 0.12 (0.599) | -6.37 (11.503)
  CD11c Dermis non lesional baseline (n=19,10) | 17.86 (7.322) | 22.97 (12.248)
  CD11c Dermis non lesional D8 (n=19,10) | 18.33 (8.971) | 20.22 (10.861)
  CD11c Dermis non lesional D8 (n=19,10) Change | 0.42 (7.613) | -2.75 (6.149)
  CD11c Dermis non lesional D29 (n=4,0) | 15.63 (10.636) | NA (NA) — no observations made
  CD11c Dermis non lesional D29 (n=4,0) Change | 0.93 (15.472) | NA (NA) — no observations made
  CD11c Dermis non lesional D85 (n=18,8) | 17.05 (5.656) | 23.73 (19.031)
  CD11c Dermis non lesional D85 (n=17,8) Change | -1.52 (7.562) | -1.23 (15.514)
  CD11c Dermis non lesional D140 (n=17,7) | 22.85 (11.189) | 15.58 (9.691)
  CD11c Dermis non lesional D140 (n=16,7) Change | 3.51 (11.162) | -11.51 (15.849)
  CD11c Dermis lesional baseline(n=19,8) | 27.14 (12.552) | 22.46 (9.700)
  CD11c Dermis lesional D8(n=11,10) | 28.85 (22.240) | 22.12 (8.669)
  CD11c Dermis lesional D8(n=11,8) Change | 3.56 (16.705) | 0.99 (8.677)
  CD11c Dermis lesional D29 (n=5,0) | 27.04 (11.509) | NA (NA) — no observations made
  CD11c Dermis lesional D29 (n=5,0) Change | -0.28 (5.403) | NA (NA) — no observations made
  CD11c Dermis lesional D85 (n=10,7) | 24.82 (13.724) | 22.59 (16.719)
  CD11c Dermis lesional D85 (n=10,6) Change | -0.09 (15.000) | 4.07 (22.288)
  CD11c Dermis lesional D140 (n=6,5) | 37.33 (21.229) | 22.59 (16.719)
  CD11c Dermis lesional D140 (n=6,4) Change | 11.30 (23.485) | 12.43 (9.210)
  CD3 Epidermis non lesional Baseline (n=19,10) | 0.37 (0.593) | 0.68 (1.151)
  CD3 Epidermis non lesional Day 8 (n=19,10) | 0.49 (0.754) | 0.34 (0.422)
  CD3 Epidermis non lesional Day 8 (n=18,10) Change | 0.14 (0.636) | -0.34 (1.091)
  CD3 Epidermis non lesional Day 29 (n=4,0) | 0.32 (0.367) | NA (NA) — no observation made
  CD3 Epidermis non lesional Day 29 (n=4,0) Change | 0.07 (0.094) | NA (NA) — no observation made
  CD3 Epidermis non lesional Day 85 (n=18,8) | 0.47 (0.660) | 0.30 (0.283)
  CD3 Epidermis non lesional Day 85 (n=17,8) Change | 0.14 (0.438) | -0.46 (1.249)
  CD3 Epidermis non lesional Day 140 (n=17,7) | 0.36 (0.470) | 0.75 (1.245)
  CD3 Epidermis non lesional Day 140 (n=16,7) Change | -0.08 (0.554) | -0.09 (2.092)
  CD3 Epidermis lesional Baseline (n=19,8) | 0.42 (0.459) | 0.49 (0.892)
  CD3 Epidermis lesional Day 8(n=11,10) | 0.55 (0.561) | 0.84 (0.913)
  CD3 Epidermis lesional Day 8(n=11,10) Change | 0.14 (0.604) | 0.11 (1.058)
  CD3 Epidermis lesional Day 29(n=5,0) | 0.28 (0.438) | NA (NA) — no observations made
  CD3 Epidermis lesional Day 29(n=5,0) Change | -0.33 (0.574) | NA (NA) — no observations made
  CD3 Epidermis lesional Day 85(n=10,7) | 0.46 (0.558) | 0.47 (0.499)
  CD3 Epidermis lesional Day 85(n=10,6) Change | 0.07 (0.672) | -0.09 (0.873)
  CD3 Epidermis lesional Day 140(n=7,5) | 0.84 (0.983) | 0.94 (0.969)
  CD3 Epidermis lesional Day 140(n=7,4) Change | 0.27 (0.843) | 0.98 (0.642)
  CD3 Dermis non lesional Baseline(n=19,10) | 9.97 (4.924) | 12.46 (7.954)
  CD3 Dermis non lesional Day 8(n=19,10) | 10.81 (5.359) | 8.66 (4.495)
  CD3 Dermis non lesional Day 8(n=18,10) Change | 0.72 (6.503) | -3.80 (5.984)
  CD3 Dermis non lesional Day 29(n=4,0) | 6.87 (1.427) | NA (NA) — no observation made
  CD3 Dermis non lesional Day 29(n=4,0) Change | -1.78 (3.096) | NA (NA) — no observaions made
  CD3 Dermis non lesional Day 85(n=18,8) | 12.71 (9.845) | 11.46 (7.900)
  CD3 Dermis non lesional Day 85(n=18,8) Change | 2.61 (8.287) | -2.09 (5.865)
  CD3 Dermis non lesional Day 140(n=17,7) | 11.80 (6.960) | 7.22 (5.823)
  CD3 Dermis non lesional Day 140(n=16,7) Change | 1.03 (5.717) | -6.15 (10.618)
  CD3 Dermis lesional Baseline(n=19,8) | 12.75 (6.934) | 11.94 (6.245)
  CD3 Dermis lesional Day 8 (n=11,10) | 14.93 (8.543) | 12.56 (8.894)
  CD3 Dermis lesional Day 8 (n=11,10) Change | 2.07 (6.576) | 1.58 (7.177)
  CD3 Dermis lesional Day 29 (n=5,0) | 13.08 (7.275) | NA (NA) — no observations made
  CD3 Dermis lesional day 29 (n=5,0) Change | 0.78 (10.054) | NA (NA) — no observations made
  CD3 Dermis lesional Day 85 (n=10,7) | 11.01 (3.615) | 14.44 (13.122)
  CD3 Dermis lesional Day 85 (n=10,6) Change | 0.46 (5.775) | 2.24 (13.351)
  CD3 Dermis lesional Day 140 (n=7,5) | 12.42 (7.600) | 14.58 (19.403)
  CD3 Dermis lesional Day 140(n=7,4) Change | 0.93 (10.179) | 6.33 (20.884)
  CD4 Epidermis non lesional Baseline (n=19,10) | 0.99 (1.400) | 1.07 (1.018)
  CD4 Epidermis non lesional Day 8 (n=19,10) | 1.20 (1.428) | 1.46 (1.639)
  CD4 Epidermis non lesional Day 8 (n=18,10) Change | 0.33 (1.287) | 0.39 (1.826)
  CD4 Epidermis non lesional Day 29 (n=4,0) | 1.43 (1.144) | NA (NA) — no observation made
  CD4 Epidermis non lesional Day 29 (n=4,0) change | -0.13 (0.922) | NA (NA) — no observations made
  CD4 Epidermis non lesional Day 85(n=18,8) | 0.69 (1.528) | 0.44 (0.360)
  CD4 Epdiermis non lesional Day 85(n=18,8) Change | -0.31 (2.239) | -0.49 (0.797)
  CD4 Epidermis non lesional Day 140(n=17,7) | 0.81 (0.742) | 0.76 (1.355)
  CD4 Epidermis non lesional Day 140(n=16,7) Change | -0.07 (1.283) | -0.04 (1.802)
  CD4 Epidermis lesional Baseline(n=19,8) | 0.95 (1.066) | 0.91 (1.204)
  CD4 Epidermis lesional Day 8(n=11,10) | 0.63 (0.725) | 0.90 (0.920)
  CD4 Epidermis lesional Day 8(n=11,8) Change | -0.46 (1.193) | -0.04 (0.680)
  CD4 Epidermis lesional Day 29(n=5,0) | 1.52 (1.927) | NA (NA) — no observation made
  CD4 Epdiermis lesional Day 29(n=5,0) Change | 0.12 (1.726) | NA (NA) — no observation made
  CD4 Epidermis lesional Day 85(n=10,7) | 0.68 (0.691) | 0.47 (0.432)
  CD4 Epidermis lesional Day 85(n=10,6) Change | -0.20 (0.847) | -0.78 (1.3489)
  CD4 Epidermis lesional Day 140(n=6,5) | 0.03 (0.082) | 0.84 (0.518)
  CD4 Epidermis lesional Day 140(n=6,4) Change | -0.61 (1.281) | -0.73 (1.473)
  CD4 Dermis non lesional Baseline(n=19,10) | 16.81 (6.868) | 19.39 (13.966)
  CD4 Dermis non lesional Day 8(n=19,10) | 17.80 (8.144) | 16.04 (10.590)
  CD4 Dermis non lesional Day 8(n=18,10) Change | 1.21 (9.816) | -3.35 (10.063)
  CD4 Dermis non lesional Day 29(n=4,0) | 15.58 (5.070) | NA (NA) — no observation made
  CD4 Dermis non lesional Day 29(n=4,0) Change | -0.88 (1.928) | NA (NA) — no observation made
  CD4 Dermis non lesional Day 85(n=18,8) Change | 19.33 (7.741) | 19.21 (10.316)
  CD4 Dermis non lesional Day 85(n=17,8) Change | 1.94 (10.126) | -2.32 (9.451)
  CD4 Dermis non lesional Day 140(n=17,7) | 21.14 (11.300) | 16.90 (10.151)
  CD4 Dermis non lesional Day 140(n=16,7) Change | 3.36 (11.994) | -2.01 (13.600)
  CD4 Dermis lesional baseline(n=19,8) | 14.28 (5.351) | 18.98 (9.361)
  CD4 Dermis lesional Day 8(n=11,10) | 17.84 (10.403) | 17.74 (9.230)
  CD4 Dermis lesional Day 8(n=11,8) Change | 2.86 (7.576) | 0.10 (10.085)
  CD4 Dermis lesional Day 29(n=5,0) | 17.12 (8.146) | NA (NA) — no observation made
  CD4 Dermis lesional Day 29(n=5,0) Change | 3.20 (4.250) | NA (NA) — no ondervation made
  CD4 Dermis lesional Day 85(n=10,7) | 17.20 (6.815) | 19.80 (12.617)
  CD4 Dermis lesional Day 85(n=10,6) Change | 3.41 (7.859) | 0.98 (10.706)
  CD4 Dermis lesional Day 140(n=6,5) | 12.81 (10.305) | 19.80 (12.617)
  CD4 Dermis lesional Day 140(n=6,4) Change | 2.58 (11.073) | -0.15 (11.300)
  CD8 Epidermis non lesional Baseline(n=19,10) | 0.20 (0.306) | 0.24 (0.420)
  CD8 Epidermis non lesional Day 8(n=19,10) | 0.40 (0.593) | 0.20 (0.340)
  CD8 Epidermis non lesional Day 8(n=18,10) Change | 0.24 (0.550) | -0.04 (0.532)
  CD8 Epidermis non lesional Day 29(n=4,0) | 0.39 (0.347) | NA (NA) — no observation made
  CD8 Epidermis non lesional Day 29(n=4,0) Change | -0.21 (0.448) | NA (NA) — no observation made
  CD8 Epidermis non lesional Day 85(n=18,8) | 0.22 (0.361) | 0.15 (0.207)
  CD8 Epidermis non lesional Day 85(n=17,8) Change | 0.00 (0.473) | -0.13 (0.354)
  CD8 Epidermis non lesional Day 140(n=17,7) | 0.16 (0.215) | 0.28 (0.351)
  CD8 Epidermis non lesional Day 140(n=16,7) Change | -0.04 (0.344) | -0.01 (0.566)
  CD8 Epidermis lesional Baseline(n=19,8) | 0.34 (0.644) | 0.14 (0.207)
  CD8 Epidermis lesional Day 8(n=11,10) | 0.43 (0.568) | 0.08 (0.140)
  CD8 Epidermis lesional Day 8(n=11,8) Change | 0.30 (0.534) | -0.11 (0.236)
  CD8 Epidermis lesional Day 29(n=5,0) | 0.20 (0.346) | NA (NA) — no observation made
  CD8 Epidermis lesional Day 29(n=5,0) Change | 0.08 (0.363) | NA (NA) — no observation made
  CD8 Epidermis lesional Day 85(n=10,7) | 0.14 (0.313) | 0.03 (0.076)
  CD8 Epidermis lesional Day 85(n=10,6) Change | -0.01 (0.356) | -0.15 (0.235)
  CD8 Epidermis lesional Day 140(n=6,5) | 0.03 (0.082) | 0.33 (0.239)
  CD8 Epidermis lesional Day 140(n=6,4) Change | -0.53 (1.129) | 0.18 (0.304)
  CD8 Dermis non lesional Baseline(n=19,10) | 5.74 (3.278) | 6.59 (3.826)
  CD8 Dermis non lesional Day 8(n=19,10) | 7.10 (5.020) | 5.50 (3.779)
  CD8 Dermis non lesional Day 8 (n=18,10) Change | 1.19 (4.798) | -1.09 (1.374)
  CD8 Dermis non lesional Day 29(n=4,0) | 8.45 (5.369) | NA (NA) — no observation made
  CD8 Dermis non lesional Day 29(n=4,0) Change | 1.80 (1.849) | NA (NA) — no observation made
  CD8 Dermis non lesional Day 85 (n=18,8) Change | 5.51 (3.725) | 7.62 (4.288)
  CD8 Dermis non lesional Day 85 (n=17,8) Change | -0.46 (2.757) | 0.35 (3.067)
  CD8 Dermis non lesional Day 140(n=17,7) Change | 4.30 (2.357) | 5.09 (3.523)
  CD8 Dermis non lesional Day 140(n=16,7) Change | -1.74 (2.726) | -2.65 (1.686)
  CD8 Dermis lesional Baseline(n=19,8) | 5.67 (2.983) | 4.63 (2.448)
  CD8 Dermis non lesional Day 8(n=11,10) | 7.55 (4.953) | 6.12 (3.847)
  CD8 Dermis non lesional Day 8(n=11,8) Change | 1.02 (5.174) | 0.88 (2.679)
  CD8 Dermis non lesional Day 29(n=5,0) | 10.14 (6.133) | NA (NA) — no observation made
  CD8 Dermis non lesional Day 29(n=5,0) Change | 2.48 (5.639) | NA (NA) — no observation made
  CD8 Dermis non lesional Day 85(n=10,7) | 7.19 (3.022) | 6.70 (6.690)
  CD8 Dermis non lesional Day 85(n=10,6) Change | 0.98 (3.556) | 1.48 (6.628)
  CD8 Dermis non lesional Day 140(n=6,5) | 7.73 (6.774) | 6.37 (10.549)
  CD8 Dermis non lesional Day 140(n=6,4) | 1.87 (7.440) | 3.57 (10.671)
  CD117 Epidermis non lesional Baseline (n=19,10) | 9.47 (5.070) | 10.99 (4.498)
  CD117 Epidermis non lesional Day 8 (n=19,10) | 10.29 (4.555) | 9.68 (3.057)
  CD117 Epidermis non lesional Day 8 (n=18,10) Chge | 0.99 (5.511) | -1.31 (2.493)
  CD117 Epidermis non lesional Day 29 (n=4,0) | 12.00 (4.578) | NA (NA) — no observationmade
  CD117 Epidermis non lesional Day 29 (n=4,0) Chge | 1.05 (2.996) | NA (NA) — no observation made
  CD117 Epidermis non lesional Day 85 (n=18,8) | 8.75 (4.492) | 9.17 (2.550)
  CD117 Epidermis non lesional Day 85 (n=17,8) Chge | -1.62 (5.338) | -1.02 (4.166)
  CD117 Epidermis non lesional Day 140 (n=17,7) | 9.89 (3.427) | 8.01 (2.744)
  CD117 Epidermis non lesional Day 140 (n=16,7) Chge | 0.023 (3.866) | -2.43 (2.234)
  CD117 Epidermis lesional baseline(n=19,8) | 7.64 (3.710) | 10.18 (3.804)
  CD117 Epidermis lesional Day 8(n=11,10) | 11.25 (5.742) | 10.84 (3.865)
  CD117 Epidermis lesional Day 8(n=11,8) Change | 2.58 (4.315) | 1.42 (5.978)
  CD117 Epidermis lesional Day 29(n=5,0) | 14.06 (4.272) | NA (NA) — no observation made
  CD117 Epidermis lesional Day 29(n=5,0) Change | 3.74 (4.844) | NA (NA) — no observation made
  CD117 Epidermis lesional Day 85(n=10,7) | 10.68 (6.160) | 8.77 (2.606)
  CD117 Epidermis lesional Day 85(n=10,6) Change | 2.10 (5.703) | -0.97 (3.885)
  CD117 Epidermis lesional Day 140(n=6,5) | 9.88 (4.399) | 8.66 (2.136)
  CD117 Epidermis lesional Day 140(n=6,4) Change | 2.41 (3.792) | -0.98 (3.444)
  CD117 Dermis non lesional Baseline (n=19,10) | 10.59 (6.616) | 10.11 (2.910)
  CD117 Dermis non lesional Day 8 (n=19,10) | 12.00 (6.370) | 9.20 (3.319)
  CD117 Dermis non lesional Day 8 (n=18,10) Change | 1.49 (5.924) | -0.91 (3.078)
  CD117 Dermis non lesional Day 29 (n=4,0) | 10.08 (2.062) | NA (NA) — no observation made
  CD117 Dermis non lesional Day 29 (n=4,0) Change | -0.47 (2.968) | NA (NA) — no observation made
  CD117 Dermis non lesional Day 85 (n=18,8) | 10.93 (6.046) | 11.18 (4.568)
  CD117 Dermis non lesional Day 85 (n=17,8) Change | -0.01 (5.750) | 0.52 (3.239)
  CD117 Dermis non lesional Day 140(n=17,7) | 12.05 (4.212) | 7.22 (2.100)
  CD117 Dermis non lesional Day 140 (n=16,7) Change | 0.69 (5.439) | -3.79 (2.284)
  CD117 Dermis lesional Baseline(n=19,8) | 9.00 (4.570) | 7.31 (2.468)
  CD117 Dermis lesional Day 8(n=11,10) | 10.15 (6.629) | 8.08 (2.743)
  CD117 Dermis lesional Day 8(n=11,8) Change | 0.60 (4.374) | 1.26 (2.890)
  CD117 Dermis lesional Day 29(n=5,0) | 12.42 (5.175) | NA (NA) — no observation made
  CD117 Dermis lesional Day 29(n=5,0) Change | 5.39 (5.412) | NA (NA) — no observation made
  CD117 Dermis lesional Day 85(n=10,7) | 11.07 (6.023) | 9.51 (2.891)
  CD117 Dermis lesional Day 85(n=10,6) Change | 2.11 (5.917) | 3.03 (2.659)
  CD117 Dermis lesional Day 140(n=6,5) | 10.92 (6.704) | 8.87 (4.017)
  CD117 Dermis lesional Day 140(n=6,4) Change | 5.12 (6.410) | 2.88 (4.907)
  Giemsa Epidermis non lesional Baseline (n=19,10) | 0.00 (0.000) | 0.00 (0.000)
  Giemsa Epidermis non lesional Day 8 (n=19,10) | 0.00 (0.000) | 0.00 (0.000)
  Giemsa Epidermis non lesional Day 8 (n=18,10) Chge | 0.00 (0.000) | 0.00 (0.000)
  Giemsa Epidermis non lesional Day 29 (n=4,0) | 0.00 (0.000) | NA (NA) — no observation made
  Giemsa Epidermis non lesional Day 29 (n=4,0) Chge | 0.00 (0.000) | NA (NA) — no observation made
  Giemsa Epidermis non lesional Day 85 (n=18,8) | 0.00 (0.000) | 0.00 (0.000)
  Giemsa Epidermis non lesional Day 85 (n=17,8) | 0.00 (0.000) | 0.00 (0.000)
  Giemsa Epidermis non lesional Day 140(n=18,8) | 0.00 (0.000) | 0.00 (0.000)
  Giemsa Epidermis non lesional Day 140(n=17,8) Chge | 0.00 (0.000) | 0.00 (0.000)
  Giemsa Epidermis lesional Baseline (n=19,8) | 0.00 (0.000) | 0.03 (0.071)
  Giemsa Epidermis lesional Day 8 (n=11,10) | 0.00 (0.000) | 0.00 (0.000)
  Giemsa Epidermis lesional Day 8 (n=11,8) Chge | 0.00 (0.000) | -0.03 (0.071)
  Giemsa Epidermis lesional Day 29(n=5,0 ) | 0.00 (0.000) | NA (NA) — no observation made
  Giemsa Epidermis lesional Day 29(n=5,0 ) Chge | 0.00 (0.000) | NA (NA) — no observation made
  Giemsa Epidermis lesional Day 85 (n=10,6) | 0.00 (0.000) | 0.00 (0.000)
  Giemsa Epidermis lesional Day 85 (n=10,5) Chge | 0.00 (0.000) | -.04 (0.089)
  Giemsa Epidermis lesional Day 140(n=6,5 ) | 0.00 (0.000) | 1.00 (2.236)
  Giemsa Epidermis lesional Day 140(n=6,4 ) Chge | 0.00 (0.000) | 1.25 (2.500)
  Giemsa Dermis non lesional Baseline (n=19,10 ) | 6.91 (4.751) | 6.80 (8.610)
  Giemsa Dermis non lesional Day 8 (n=19,10 ) | 5.51 (4.142) | 4.47 (4.529)
  Giemsa Dermis non lesional Day 8 (n=18,10 ) Chge | -1.33 (5.141) | -2.33 (4.750)
  Giemsa Dermis non lesional Day 29 (n=4,0 ) | 3.88 (1.876) | NA (NA) — no observation made
  Giemsa Dermis non lesional Day 29 (n=4,0 ) Chge | -1.62 (1.811) | NA (NA) — no observation made
  Giemsa Dermis non lesional Day 85 (n=18,8 ) | 4.75 (3.397) | 5.28 (4.906)
  Giemsa Dermis non lesional Day 85 (n=17,8 ) Chge | -2.34 (3.618) | -2.16 (6.705)
  Giemsa Dermis non lesional Day 140 (n=18,10 ) | 6.69 (5.409) | 3.12 (3.120)
  Giemsa Dermis non lesional Day 140 (n=18,10 ) Chge | -1.35 (5.078) | -4.86 (7.348)
  Giemsa Dermis lesional Baseline(n=19,8 ) | 8.29 (5.189) | 4.79 (5.931)
  Giemsa Dermis lesional Day 8(n=11,10 ) | 6.71 (4.309) | 4.80 (4.512)
  Giemsa Dermis lesional Day 8(n=11,8 ) Chge | -1.75 (6.143) | 0.18 (3.394)
  Giemsa Dermis lesional Day 29(n=5,0 ) | 8.09 (11.851) | NA (NA) — no observation made
  Giemsa Dermis lesional Day 29(n=5,0 ) Chge | 2.57 (12.812) | NA (NA) — no observation made
  Giemsa Dermis lesional Day 85(n=10,6 ) | 5.96 (2.589) | 10.30 (15.647)
  Giemsa Dermis lesional Day 85 (n=10,5 ) Chge | -1.56 (7.155) | 6.36 (9.563)
  Giemsa Dermis lesional Day 140(n=6,5 ) | 7.57 (2.589) | 9.44 (10.468)
  Giemsa Dermis lesional Day 140 (n=6,4 ) Chge | -1.20 (7.929) | 4.50 (5.073)
  H&E Epidermis non lesional Baseline(n=19,10 ) | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis non lesional day 8(n=19,10 ) | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis non lesional Day 8(n=18,10 ) Chge | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis non lesional Day 29(n=4,0 ) | 0.00 (0.000) | NA (NA) — no observation made
  H&E Epidermis non lesional Day 29(n=4,0 ) Chge | 0.00 (0.000) | NA (NA) — no observation made
  H&E Epidermis non lesional Day 85(n=17,8 ) | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis non lesional Day 85(n=16,8 ) Chge | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis non lesional Day 140 (n=17,7 ) | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis non lesional Day 140 (n=16,7 ) Chge | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis lesional Baseline(n=19,8 ) | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis lesional Day 8(n=11,10 ) | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis lesional Day 8(n=11,8 ) Chge | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis lesional Day 29(n=5,0 ) | 0.00 (0.000) | NA (NA) — no observation made
  H&E Epidermis lesional Day 29(n=5,0 ) Chge | 0.00 (0.000) | NA (NA) — no observation made
  H&E Epidermis lesional Day 85(n=10,6 ) | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis lesional Day 85(n=10,5 ) Chge | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis lesional Day 140(n=6,5 ) | 0.00 (0.000) | 0.00 (0.000)
  H&E Epidermis lesional Day 140(n=6,4 ) Chge | 0.00 (0.000) | 0.00 (0.000)
  H&E Dermis non lesional Baseline(n=19,10 ) | 0.00 (0.000) | 0.00 (0.000)
  H&E Dermis non lesional Day 8(n=19,10 ) | 0.01 (0.046) | 0.02 (0.063)
  H&E Dermis non lesional Day 8(n=18,10 ) Chge | 0.01 (0.047) | 0.02 (0.063)
  H&E Dermis non lesional Day 29(n=4,0 ) | 0.00 (0.000) | NA (NA) — no observation made
  H&E Dermis non lesional Day 29(n=4,0 ) Chge | 0.00 (0.000) | NA (NA) — no observation made
  H&E Dermis non lesional Day 85(n=17,8) | 0.00 (0.000) | 0.00 (0.000)
  H&E Dermis non lesional Day 85(n=16,8 ) Chge | 0.00 (0.000) | 0.00 (0.000)
  H&E Dermis non lesional Day 140(n=17,7 ) | 0.00 (0.000) | 0.03 (0.076)
  H&E Dermis non lesional Day 140(n=16,7 ) Chge | 0.00 (0.000) | 0.03 (0.076)
  H&E Dermis lesional Baseline(n=19,8 ) | 0.02 (0.071) | 0.03 (0.071)
  H&E Dermis lesional Day 8(n=11,10 ) | 0.05 (0.129) | 0.00 (0.000)
  H&E Dermis lesional Day 8(n=11,8 ) Chge | 0.03 (0.159) | -0.03 (0.071)
  H&E Dermis lesional Day 29(n=5,0 ) | 0.00 (0.000) | NA (NA) — no observation made
  H&E Dermis lesional Day 29(n=5,0 ) Chge | 0.00 (0.000) | NA (NA) — no observation made
  H&E Dermis lesional Day 85(n=10,6 ) | 0.00 (0.000) | 0.03 (0.082)
  H&E Dermis lesional Day 85(n=10,5 ) Chge | 0.00 (0.000) | 0.04 (0.089)
  H&E Dermis lesional Day 140(n=6,5 ) | 0.00 (0.000) | 0.00 (0.000)
  H&E Dermis lesional Day 140(n=6,4 ) Chge | 0.00 (0.000) | 0.00 (0.000)
  Tryptase Epidermis non lesional Baseline (n=19,10) | 0.00 (0.000) | 0.00 (0.000)
  Tryptase Epidermis non lesional Day 8 (n=19,10) | 0.02 (0.092) | 0.00 (0.000)
  Tryptase Epidermis non lesional Day 8(n=18,10) Chg | 0.02 (0.094) | 0.00 (0.000)
  Tryptase Epidermis non lesional Day 29 (n=4,0) | 0.00 (0.000) | NA (NA) — no observation made
  Tryptase Epidermis non lesional Day 29 (n=4,0) Chg | 0.00 (0.000) | NA (NA) — no observation made
  Tryptase Epidermis non lesional Day 85 (n=18,8) | 0.03 (0.103) | 0.00 (0.000)
  Tryptase Epidermis non lesional Day 85(n=17,8) Chg | 0.04 (0.100) | 0.00 (0.000)
  Tryptase Epidermis non lesional Day 140 (n=17,7) | 0.02 (0.097) | 0.00 (0.000)
  Tryptase Epidermis non lesional Day140(n=16,7) Chg | 0.03 (0.100) | 0.00 (0.000)
  Tryptase Epidermis lesional Baseline (n=19,8) | 0.01 (0.046) | 0.08 (0.149)
  Tryptase Epidermis lesional day 8 (n=11,10) | 0.33 (1.085) | 0.10 (0.316)
  Tryptase Epidermis lesional Day 8 (n=11,8) Chg | 0.31 (1.093) | 0.05 (0.334)
  Tryptase Epidermis lesional Day 29 (n=5,0) | 0.12 (0.268) | NA (NA) — no observation made
  Tryptase Epidermis lesional Day 29 (n=5,0) Chg | 0.08 (0.179) | NA (NA) — no observation made
  Tryptase Epidermis lesional Day 85(n=10,7) | 0.00 (0.000) | 0.00 (0.000)
  Tryptase Epidermis lesional Day 85(n=10,6) Chg | -0.02 (0.063) | -0.10 (0.167)
  Tryptase Epidermis lesional Day 140 (n=7,5) | 0.00 (0.000) | 0.00 (0.000)
  Tryptase Epidermis lesional Day 140 (n=7,4) Chg | -0.03 (0.076) | -0.10 (0.200)
  Tryptase Dermis non lesional Baseline (n=19,10) | 6.55 (3.988) | 7.20 (3.045)
  Tryptase Dermis non lesional Day 8 (n=19,10) | 7.14 (4.479) | 8.37 (2.305)
  Tryptase Dermis non lesional Day 8 (n=18,10) Chg | 1.14 (2.989) | 1.17 (3.030)
  Tryptase Dermis non lesional Day 29 (n=4,0) | 8.22 (4.981) | NA (NA) — no observation made
  Tryptase Dermis non lesional Day 29 (n=4,0) Chg | 0.67 (4.816) | NA (NA) — no observation made
  Tryptase Dermis non lesional Day 85 (n=18,8) | 7.66 (4.076) | 8.33 (3.547)
  Tryptase Dermis non lesional Day 85 (n=17,8) Chg | 0.54 (3.753) | 1.35 (3.839)
  Tryptase Dermis non lesional Day 140 (n=17,7) | 7.77 (4.296) | 6.95 (1.812)
  Tryptase Dermis non lesional Day 140 (n=16,7) Chg | 1.27 (3.599) | -0.62 (3.002)
  Tryptase Dermis lesional Baseline (n=19,8) | 6.08 (3.764) | 6.41 (2.658)
  Tryptase Dermis lesional Day 8 (n=11,10) | 7.19 (3.618) | 6.99 (3.451)
  Tryptase Dermis lesional Day 8 (n=11,8) Chg | 0.71 (2.809) | 0.88 (2.998)
  Tryptase Dermis lesional Day 29(n=5,0) | 10.20 (4.658) | NA (NA) — no observation made
  Tryptase Dermis lesional Day 29(n=5,0) Chg | 3.80 (3.023) | NA (NA) — no observation made
  Tryptase Dermis lesional Day 85(n=10,7) | 6.76 (3.082) | 6.93 (3.135)
  Tryptase Dermis lesional Day 85(n=10,6) Chg | 0.39 (4.141) | 1.67 (2.047)
  Tryptase Dermis lesional Day 140(n=7,5) | 6.59 (6.335) | 6.79 (1.635)
  Tryptase Dermis lesional Day 140(n=7,4) Chg | 2.68 (6.641) | 1.97 (2.049)

6. Secondary Outcome: Observed Values From Baseline Through End of Study of Serum Chemkines or Histamine in Peripheral Blood Cells by Parameter, Treatment and Visit
Time Frame: Baseline through Day 85
Population: All subjects who received at least one dose of study drug and had evaluable pharmacodynamic (PD) data were included in the PD data analysis.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
ug/mL
  Chemokine CCR3 Baseline (n=19,10) | 2.9669 (2.31825) | 3.0394 (2.38102)
  Chemokine CCR3 Day 2 (n=20, 10) | 2.8190 (2.94786) | 3.3035 (3.52023)
  Chemokine CCR3 Day 8 (n=20,10) | 2.5597 (2.22009) | 2.2742 (1.58648)
  Chemokine CCR3 Day 15 (n=19,8) | 2.2711 (1.98781) | 2.0216 (1.46346)
  Chemokine CCR3 Day 29 (n=20,9) | 2.5869 (2.31661) | 2.2826 (1.56237)
  Chemokine CCR3 Day 85 (n=17,8) | 2.5178 (1.93931) | 1.8724 (1.16171)
  Chemokine CCR3 Day 140 (n=18,10) | 2.022 (2.44218) | 2.4060 (1.85351)
  Chemokine CXCR3/IP-10 Baseline (n=19,10) | 0.1020 (0.07807) | 0.0638 (0.07208)
  Chemokine CXCR3/IP-10 Day 2 (n=20,9) | 0.0836 (0.06630) | 0.0621 (0.06496)
  Chemokine CXCR3/IP-10 Day 8 (n=19,8) | 0.0910 (0.07704) | 0.0772 (0.05990)
  Chemokine CXCR3/IP-10 Day 15 (n=19,7) | 0.0883 (0.06303) | 0.0546 (0.02550)
  Chemokine CXCR3/IP-10 Day 29 (n=20,9) | 0.0881 (0.07624) | 0.0601 (0.04219)
  Chemokine CXCR3/IP-10 Day 85 (n=17,8) | 0.0714 (0.03079) | 0.0430 (0.02910)
  Chemokine CXCR3/IP-10 Day 140 (n=18,9) | 0.0864 (0.07319) | 0.0859 (0.07489)
  Histamine Baseline (n=19,10) | 5.0526 (2.06757) | 5.2000 (1.13529)
  Histamine Day 2 (n=20,10) | 4.1500 (1.6111) | 5.0000 (1.76383)
  Histamine Day 8 (n=20,10) | 4.5000 (2.01311) | 5.4000 (2.01108)
  Histamine Day 15 (n=19,8) | 4.5789 (1.64370) | 4.7500 (1.83225)
  Histamine Day 29 (n=20,9) | 5.1500 (2.20705) | 4.7778 (3.38296)
  Histamine Day 85 (n=17,8) | 5.8235 (1.50977) | 5.0000 (1.30931)
  Histamine Day 140 (n=18,10) | 4.8333 (2.64019) | 5.7000 (1.76698)
  Chemokine ICAM-1 Baseline (n=19,10) | 0.4858 (0.09955) | 0.5191 (0.14846)
  Chemokine ICAM-1 Day 2 (n=20,10) | 0.4468 (0.07872) | 0.4975 (0.14406)
  Chemokine ICAM-1 Day 8 (n=20,10) | 0.4967 (0.12551) | 0.4728 (0.15713)
  Chemokine ICAM-1 Day 15 (n=19,8) | 0.4788 (0.12577) | 0.4709 (0.11789)
  Chemokine ICAM-1 Day 29 (n=20,9) | 0.4633 (0.10172) | 0.4704 (0.11356)
  Chemokine ICAM-1 Day 85 ( n= 17,8) | 0.4314 (0.10424) | 0.4037 (0.05599)
  Chemokine ICAM-1 Day 140 ( n=15,10) | 0.4314 (0.10921) | 0.4918 (0.15250)

7. Secondary Outcome: Observed Values and Change From Baseline in Peripheral Blood Cell Subsets (FACS Parameters) at Week 12 (Day 85) by Treatment (PD Analysis Set) Measured as % Out of Leukocytes.
Description: Fluorescence-activated cell sorting (FACS) is a specialized type of flow cytometry that provides a method for sorting a heterogeneous mixture of biological cells into two or more containers, one cell at a time, based upon the specific light scattering and fluorescent characteristics of each cell. (FACS) provides fast, objective and quantitative recording of fluorescent signals from individual cells as well as physical separation of cells of particular interest. A wide range of fluorophores can be used as labels in flow cytometry. Fluorophores are typically attached to an antibody that recognizes a target feature on or in the cell; they may also be attached to a chemical entity with affinity for the cell membrane or another cellular structure. Each fluorophore has a characteristic peak excitation and emission wavelength.
Time Frame: Baseline through Day 85
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: % out of leukocytes
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
% out of leukocytes
  Basophils D1 (n=19,10) Units | 0.23 (0.132) | 0.36 (0.482)
  Basophils D85 (n=7,5) Units | 0.47 (0.215) | 0.40 (0.451)
  Basophils chge (n=7,5) Units | 0.22 (0.268) | -0.06 (0.176)
  CD19+ B cells bound IgE D1 (n=8,8) | 4.53 (5.001) | 15.19 (22.609)
  CD19+ B cells bound IgE D85(n=5,7) | 7.32 (7.579) | 25.66 (26.485)
  CD19+ B cells bound IgE chge (n=5,7 | 1.46 (3.545) | 12.53 (21.725)
  CD19+ B cells D1 (n=10,9) | 3.57 (2.298) | 2.5 (1.247)
  CD19+ B cells D85 (n=7,7) | 3.84 (1.595) | 3.25 (2.007)
  CD19+ B cells Chge (n=7,7) | 0.31 (1.377) | 0.73 (0.805)
  Dendritic cells D1 (n=10,7) | 0.37 (0.196) | 0.24 (0.140)
  Dendritic cells D85 (n=8,5) | 0.37 (0.231) | 0.27 (0.210)
  Dendritic cells Chge (n=7,5) | 0.02 (0.272) | -0.02 (0.182)

8. Secondary Outcome: Observed Values and Change From Baseline in Peripheral Blood Cell Subsets (FACS Parameters) at Week 12 (Day 85) by Treatment (PD Analysis Set) Measured in Fluorescence Units.
Description: as for outcome 7
Time Frame: Baseline through Day 85
Population: All subjects who received at least one dose of study drug and had evaluable pharmacodynamic (PD) data were included in the PD data analysis.• FACS parameters: FceRI expression on basophils and IgE bound, FceR2 expression on B cells and IgE bound, and FceRI expression on dendritic cells
Measure: Mean (Standard Deviation); unit: Flourescence units
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
Flourescence units
  Basophils with FcεR1 exp D1 (n=11,8) | 292391 (135848) | 312038 (147037)
  Basophils with FcεR1 exp D85 (n=7,5) | 79457 (29333) | 291000 (108028)
  Basophils with FcεR1 expression Chge (n=6,5) | -243700 (118883) | -38260 (60085)
  Basophils with bound IgE D 1 (n=11,7) | 149656 (112936) | 236071 (89043)
  Basophils with bound IgE D85 (n=7,5) | 9554 (6214) | 212620 (109645)
  Basophils with bound IgE Chge (n=6,5) | -178487 (103456) | -12680 (59998)
  CD19+ B cells with FcεR2 exp D1 (n=10,9) | 59040 (42446) | 59700 (27171)
  CD19+ B cells with FcεR2 exp D85 (n=7,7) | 59429 (55980) | 49243 (33460)
  CD19+ B cells with FcεR2 exp chge (n=7,7) | 12814 (32631) | 3986 (16779)
  Dendritic cells with FcεR1 expr D1 (n=10,7) | 40880 (17191) | 43029 (12363)
  Dendritic cells with FcεR1 expr D85 (n=6,5) | 38283 (5768) | 36962 (18562)
  Dendritic cells with FcεR1 expr Chge (n=5,5) | -10100 (16887) | -516 (5925)

9. Secondary Outcome: Comparison of Baseline PD Parameters Between Healthy Volunteers and Urticaria Patients by Skin Layer Pharmacodynamic Analysis Set
Description: The # positive cell values are average of cell numbers derived from counting 5 consecutive microscopic fields. Area counted is 5x 0.196 mm2
Time Frame: Baseline
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: # positive cells
Groups:
- Healthy Subjects: Baseline Value, healthy volunteers, no treatment applied
- Urticaria Patients: All patients for study at baseline
Arm/Group | Healthy Subjects | Urticaria Patients
Number analyzed (Participants) | 10 | 30
# positive cells
  CD11c Epidermis ( n= 10,29) | 1.1600 (1.13058) | 1.1241 (0.92944)
  CD11c Dermis (n=10,29) | 14.6400 (9.31083) | 19.6207 (9.42260)
  CD11c All skin layers (n=20,58) | 7.9000 (9.45983) | 10.3724 (11.44855)
  CD 3 Epidermis (n=10,29) | 0.1600 (0.26331) | 0.4759 (0.82046)
  Cd 3 Dermis (n=10,29) | 10.1600 (9.00311) | 10.8276 (6.11385)
  CD 3 All Skin Layers (n=20,58) | 5.1600 (8.04634) | 5.6517 (6.77879)
  CD 4 Epidermis (n=10,29) | 1.0250 (1.75804) | 1.0207 (1.26297)
  CD 4 Dermis (n=10,29) | 15.7750 (10.06565) | 17.7000 (9.72481)
  CD 4 All Skin Layers (n=20,58) | 8.4000 (10.33004) | 9.3603 (10.86324)
  CD 8 Epidermis (n=10,29) | 0.0600 (0.13499) | 0.2138 (0.34197)
  CD 8 Dermis (n=10,29) | 5.9083 (4.07998) | 6.0322 (3.43255)
  CD 8 All Skin Layers (n=20,58) | 2.9842 (4.11029) | 3.1230 (3.80226)
  CD 117 Epidermis (n=10,29) | 10.1600 (3.80386) | 9.9931 (4.85502)
  CD 117 Dermis (n=10,29) | 8.2200 (2.44849) | 10.4241 (5.56025)
  CD 117 All Skin Layers (n=20,58) | 9.1900 (3.26865) | 10.2086 (5.17814)
  Fc epsilon receptor I Epidermis (n=10,29) | 4.9800 (2.02309) | 6.0776 (3.12906)
  Fc epsilon receptor I Dermis (n=10,29) | 14.2000 (6.76133) | 19.4500 (8.21582)
  Fc epsilon receptor I All Skin Layers (n=20,58) | 9.5900 (6.77968) | 12.7638 (9.13548)
  Giemsa Epidermis (n=10,29) | 0.0000 (0.00000) | 0.0000 (0.00000)
  Giemsa Dermis (n=10,29) | 4.8000 (5.62929) | 6.8690 (6.19228)
  Giemsa All Skin Layers (n=20,58) | 2.4000 (4.59061) | 3.4345 (5.55324)
  Haematoxylin + Eosin Epidermis (n=10,29) | 0.0000 (0.00000) | 0.0000 (0.00000)
  Haematoxylin + Eosin Dermis (n=10,29) | 0.0000 (0.00000) | 0.0000 (0.00000)
  Haematoxylin + Eosin All Skin Layers (n=20,58) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IgE Epidermis (n=10,29) | 0.0800 (0.13984) | 1.0603 (2.30385)
  IgE Dermis (n=10,29) | 8.7600 (5.92231) | 14.7776 (9.84503)
  IgE All Skin layers (n=20,58) | 4.4200 (6.03739) | 7.9190 (9.90380)
  IgE + CD 11c Epidermis (n=10,28) | 0.0000 (0.00000) | 0.0357 (0.12237)
  IgE + CD 11c Dermis (n=10,29) | 0.9150 (1.29401) | 1.0115 (1.05290)
  IgE+CD 11c All Layers (n=20,57) | 0.4575 (1.00672) | 0.5322 (0.89651)
  IgE + Tryptase Epidermis (n=10,28) | 0.0000 (0.00000) | 0.0000 (0.00000)
  IgE + Tryptase Dermis (n=10,29) | 1.3000 (1.01215) | 0.8713 (0.79919)
  IgE + Tryptase All Skin Layers (n=20,57) | 0.6500 (0.96437) | 0.4433 (0.71586)
  Tryptase Epidermis (n=10,29) | 0.0000 (0.00000) | 0.0000 (0.00000)
  Tryptase Dermis (n=10,29) | 6.6400 (3.53371) | 6.7741 (3.64713)
  Tryptase All Skin Layers (n=20,58) | 3.3200 (4.18539) | 3.3871 (4.26704)

10. Secondary Outcome: Serum Levels of Omalizumab
Description: Serum concentrations (ng/mL) of omalizumab by visit after the administration of omalizumab 300 mg every 4 weeks
Time Frame: Baseline through Day 85
Population: PK analysis set which included all subjects who received at least one dose of study drug and had evaluable IGE025 concentrations.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IGE025
Number analyzed (Participants) | 20
ng/mL
  Day 1 | 0.0 (0.00)
  Day 2 | 13400 (4690)
  Day 8 | 30100 (7800)
  Day 29 | 17000 (5500)
  Day 57 | 25000 (8640)
  Day 85 | 28800 (11400)

11. Secondary Outcome: Mean (SD) Serum Total IgE Concentration From Baseline by Visit
Time Frame: Baseline through Day 85
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
ng/mL
  Day 1 Mean (n=20,10) | 1037 (2474) | 442 (580.7)
  Day 2 Mean (20,10) | 1152 (2539) | 447 (587.5)
  Day 8 Mean (n=20,10) | 1970 (2992) | 449 (593.1)
  Day 29 Mean (n=20,9) | 2160 (2688) | 462 (628.7)
  Day 57 Mean (n=19,8) | 2430 (3343) | 490 (648.0)
  Day 85 Mean (n=17,8) | 2222 (2931) | 475 (616.8)

12. Secondary Outcome: Mean (SD) Serum Total IgE % Change From Baseline by Visit
Time Frame: Baseline through Day 85
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
Percent Change from Baseline
  Day 2 % Change (n=19,10) | 27.1 (20.08) | 0.2 (5.13)
  Day 8 % Change (n=19,10) | 174.7 (84.93) | -1.5 (9.13)
  Day 29 % Change (n=19,9) | 247.2 (121.81) | -4.0 (12.17)
  Day 57 % Change (n=18,8) | 247.8 (134.10) | -4.4 (18.59)
  Day 85 % Change (n=16,8) | 244.8 (138.28) | -6.9 (24.10)

13. Secondary Outcome: Mean (SD) Serum Free IgE Concentration From Baseline by Visit
Time Frame: Baseline through Day 85
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
ng/mL
  Day 1 Mean (n=20,10) | 1037 (2474) | 442 (580.69)
  Day 2 Mean (n= 20,9) | 26.8 (34.27) | 111.5 (60.75)
  Day 8 Mean (n=20,10) | 24.306 (29.7698) | 112.169 (58.6525)
  Day 29 Mean (n=20,9) | 41.506 (40.5322) | 107.881 (60.1708)
  Day 57 Mean (n=19,8) | 38.502 (39.5567) | 122.318 (51.1087)
  Day 85 Mean (n=17,8) | 35.776 (41.5426) | 120.978 (50.6692)

14. Secondary Outcome: Mean (SD) Serum Free IgE % Change From Baseline by Visit
Time Frame: Baseline through Day 85
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
% change
  Day 2 % Change (n=19,9) | -96.166 (2.9216) | -60.475 (17.9330)
  Day 8 % Change (n=20,10) | -96.446 (2.0162) | -60.804 (15.8379)
  Day 29 % Change (n=19,9) | -93.363 (3.5975) | -61.456 (17.2340)
  Day 57 % Change (n=18,8) | -94.460 (3.0681) | -61.270 (18.6447)
  Day 85 % Change (n=16,8) | -94.750 (3.420) | -61.906 (17.7819)

15. Secondary Outcome: Summary Statistics of Observed Values and Absolute Change From Baseline in Specific IgE Against Allergens and Bacterial Antigens by Parameter, Treatment and Visit
Time Frame: Baseline through Day 140
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 20 | 10
IU/mL
  Alternaria alternara Baseline (n= 0, 1) | NA (NA) — Specific IgE not observed | 0.1360 (NA) — one patient only tested positive
  Alternaria alternara Day 140 (n= 0,1) | NA (NA) — Specific IgE not observed | 0.1140 (NA) — one patient only tested positive
  Artemisia vulgaris (Mugwort) Baseline (n=1,1) | 0.2730 (NA) — one patient only tested positive | 1.4800 (NA) — one patient only tested positive
  Artemisia vulgaris (Mugwort) Day 140( n=0,1) | NA (NA) — Specific IgE not observed | 1.9100 (NA) — one patient only tested positive
  Cat dander Basseline (n=3,1) | 17.9677 (22.73833) | 0.6980 (NA) — one patient only tested positive
  Cat dander Day 140 (n=2,1) | 21.0100 (26.14881) | 0.8980 (NA) — one patient only tested positive
  Common silver Birch Baseline (n=6,3) | 12.3640 (19.48667) | 12.3767 (11.22609)
  Common silver Birch Day 140 (n=4,3) | 4.4890 (6.15938) | 14.8600 (16.58164)
  Dog dander Baseline (n=2,1) | 26.7720 (37.09199) | 0.5120 (NA) — one patient only tested positive
  Dog dander Day 140 (n=1,1) | 50.1000 (NA) — one patient only tested positive | 0.6690 (NA) — one patient only tested positive
  Dermatophagoides farinae Baseline (n=3,1) | 3.3333 (3.39883) | 0.4340 (NA) — one patient only tested positive
  Dermatophagoides farinae Day 140 (n=2,1) | 5.3200 (0.89095) | 0.4970 (NA) — one patient only tested positive
  Dermatophagoides pteronyssinus Baseline (n=5,1) | 2.1250 (1.46791) | 0.4550 (NA) — one patient only tested positive
  Dermatophagoides pteronyssinus Day 140(n=4,1) | 5.2463 (3.72052) | 0.5170 (NA) — one patient only tested positive
  Grey Alder (t2) Baseline (n=4,3) | 15.7650 (20.03961) | 10.9533 (10.92027)
  Grey Alder (t2) Day 140(n=3,3) | 4.4900 (5.16654) | 13.0533 (15.24029)
  German Cockroach Baseline (n=4,2) | 0.8605 (0.93609) | 0.4425 (0.62579)
  German Cockroach Day 140 (n=4,2) | 3.0263 (2.87190) | 0.4705 (0.66539)
  Hazelnut Baseline (n=3,3) | 8.9627 (14.49722) | 7.3267 (8.28160)
  Hazelnut Day 140 (n=2,3) | 1.4450 (1.50977) | 8.9927 (10.59244)
  Olive (black, fresh) Baseline (n=4,1) | 0.0890 (0.17800) | 0.0000 (NA) — one patient only tested positive
  Olive (black, fresh) Day 140 (n=3,1) | 0.1037 (0.17956) | 0.0000 (NA) — one patient only tested positive
  Platanus acerifolia Baseline (n=1,1) | 0.1210 (NA) — one patient only tested positive | 3.7100 (NA) — one patient only tested positive
  Platanus acerifolia Day 140 (n=0,1) | 0.0000 (NA) — one patient only tested positive | 4.8300 (NA) — one patient only tested positive
  Parietaria judaica Baseline(n=0,1) | 0.0000 (NA) — one patient only tested positive | 1.4900 (NA) — one patient only tested positive
  Parietaria judaica Day 140 (n=0,1) | 0.0000 (NA) — one patient only tested positive | 2.0000 (NA) — one patient only tested positive
  Staphylococcal enterotoxin A Baseline (n=20,10) | 0.7264 (3.07821) | 0.0741 (0.13580)
  Staphylococcal enterotoxin A Day 140 (n=18,10) | 1.6161 (4.39936) | 0.1077 (0.15294)
  Staphylococcal enterotoxin C Baseline (n=20,10) | 0.8976 (3.02621) | 0.1626 (0.27226)
  Staphylococcal enterotoxin C Day 140 (n=18,10) | 2.1089 (4.19834) | 0.1922 (0.28071)
  Staphylococcal enterotoxin TSST Baseline (n=20,10) | 0.5390 (1.02581) | 0.1537 (0.23902)
  Staphylococcal enterotoxin TSST Day 140 (n=18,10) | 0.8402 (1.05356) | 0.1468 (0.22155)
  Alternaria alternara Absolute Change (n = 0,1) | NA (NA) — Specific IgE not observed | -0.0220 (NA) — only 1 observation
  Artemisia vulgaris Absolute Change (n = 0,1) | NA (NA) — Specific IgE not observed | 0.4300 (NA) — only 1 observation
  Cat dander Absolute Change (n = 2,1) | -1.1315 (4.33951) | 0.2000 (NA) — only 1 observation
  Common Silver Birch Absolute Change (n = 4,3) | -10.2145 (26.47094) | 2.4833 (5.63479)
  Dog dander Absolute Change (n = 1,1) | -2.9000 (NA) — only 1 observation | 0.1570 (NA) — only 1 observation
  Dermatophagoides farinae Absolute Change(n=2,1) | 3.9350 (1.46371) | 0.0630 (NA) — only 1 observation
  Dermatophagoides pteronyssinus Abs Chge (n=4,1) | 3.6800 (3.05938) | 0.0620 (NA) — only 1 observation
  Grey Alder Absolute Change(n=3,3) | -12.6300 (27.47614) | 2.1000 (4.50900)
  German Cockroach Absolute Change(n=4,2) | 2.1658 (2.03436) | 0.0280 (0.03960)
  Hazelnut Absolute Change(n=2,3) | -11.83000 (18.15850) | 1.6660 (2.47183)
  Olive (black, fresh) Absolute Change(n=3,1) | -0.0150 (0.02598) | 0.0000 (NA) — only 1 observation
  Platanus acerifolia Absolute Change(n=0,1) | NA (NA) — Specific IgE not observed | 1.1200 (NA) — only 1 observation
  Parietaria judaica Absolute Change(n=0,1) | NA (NA) — Specific IgE not observed | 0.5100 (NA) — only 1 observation
  Staphylococcal enterotoxin A Abs chge (n=18,10) | 0.8090 (2.63582) | 0.0336 (0.09116)
  Staphylococcal enterotoxin C Abs chge (n=18,10) | 1.1116 (2.26524) | 0.0296 (0.06545)
  Staphylococcal enterotoxin TSST Abs chge(n=18,10) | 0.2608 (0.72963) | -0.0069 (0.15669)

16. Secondary Outcome: Change From Baseline in Urticaria Activity Score (UAS7)
Description: Efficacy was assessed by the urticaria activity score (UAS). UAS was completed each morning and evening on a daily basis to record patient symptoms of itch and hives via an electronic diary. The UAS is a composite eDiary-recorded score with numeric severity intensity ratings on a scale of 0-3 (0 = none to 3 = intense/severe) for 1) the number of wheals (hives); and 2) the intensity of the itch. The daily UAS is the average of the morning and evening scores and the UAS7 is the sum of the daily UAS scores over 7 days.UAS7 score: The sum of the daily UAS scores over 7 days. Range: 0-42. If fewer than 7 but at least 4 daily values were non-missing, the remaining values were imputed to be the average. This is equivalent to multiplying the average of the non missing values by 7. UAS7 score: The sum of the daily UAS scores over 7 days. Range: 0-42. A higher score indicates worse disease. A negative change score (Week 12 score minus Baseline score) indicates improvement.
Time Frame: Baseline, Day 85
Population: Efficacy analysis set which included all randomized patients who received at least one dose of study drug and had post-randomization efficacy data. If the Week 12 value was missing, it was imputed as the last available UAS7 value (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 17 | 8
units on a scale | -23.1 (12.94) [-28.5 to -17.6] | -8.1 (14.45) [-17.8 to 1.5]

17. Secondary Outcome: Likert Scale-Physician's and Patients In-clinic Global Assessment by Treatment
Description: The investigator or the person he or she designated and the patient provided scoring of the patient's global assessment of symptoms (urticaria lesions (hives) and pruritus) reflective of the patient's condition over the 12 hours prior to the visit (0 = no symptoms, 1 = mild, 2 = moderate 3 = severe
Time Frame: Baseline, Day 85
Population: Efficacy analysis set which included all randomized patients who received at least one dose of study drug and had post-randomization efficacy data
Measure: Mean (Standard Deviation); unit: score
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 17 | 8
score
  Physicians Baseline (n=17,9) | 2.0 (0.87) | 2.2 (0.83)
  Physicians Week 12, (day 85) (n=17,8) | 0.8 (1.01) | 2.0 (1.31)
  Patients Baseline (n=17,9) | 2.4 (0.87) | 2.4 (0.53)
  Patients Week 12, (day 85) (n=17,8) | 0.9 (1.05) | 1.9 (0.99)

18. Secondary Outcome: Percentage of Angioedema-free Days Weeks 4 Through 12 by Treatment
Time Frame: Day 29 to Day 85
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 17 | 8
Percentage of days | 90.9 (22.83) [87.8 to 94.0] | 70.5 (28.50) [64.9 to 76.1]

19. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) by Treatment
Description: The DLQI is a 10-item dermatology-specific health-related quality of life measure. Patients rated their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives. An overall score was calculated as well as for the following domains: Symptoms and Feelings, Daily Activities, Leisure, Work and School, Personal Relationships, Treatment.Negative score shows positive efficacy. Meaning of DLQI Scores 0-1 = no effect at all on patient's life 2-5 = small effect on patient's life 6-10 = moderate effect on patient's life 11-20 = very large effect on patient's life 21-30 = extremely large effect on patient's life. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30.
Time Frame: Baseline through Day 85
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 16 | 8
Score | -10.19 (8.159) | -3.13 (7.180)

20. Secondary Outcome: Skindex-29 by Treatment
Description: The Skindex-29 is a validated 29-item instrument to measure the effects of skin disease on patients' quality of life.Results are reported as 3 scale scores (functioning, emotions and symptoms) and a composite score (average scale score). The domain scores and the overall score are expressed on a 100-point scale, with higher scores indicating a lower level of quality of life. The cuttoff values for each category are noted below. Symtoms; 39 mild, 42 moderate,52 severe. Emotions; 24 mild, 35 moderate, 39 severe. Functioning: 21 mild, 32 moderate, 37 severe. Overal Score: 25 mild, 32 moderate, 44 severe.
Time Frame: Baseline and Day 85
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 16 | 8
Score
  Baseline (n= 16,9) | 17.98 (7.807) | 21.67 (9.068)
  Day 85 (n=16,8) | 6.17 (7.119) | 22.63 (10.276)

21. Secondary Outcome: Chronic Urticaria Quality of Life Questionnaire (Cu-Q2OL) by Treatment
Description: The Cu-Q2OL is a 23-item CIU-specific health-related quality of life questionnaire. Patients rated their CIU symptoms and the impact of their CIU on various aspects of their lives. An overall score was calculated as well for the following domains: pruritus, swelling, impact on life activities, sleep problems, limits, and looks. Zero is the minmum score and 100 the maximum score. The higher score correlates to more disease activity.
Time Frame: Baseline and Day 85
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score
Arm/Group | IGE025 | Placebo IGE025
Number analyzed (Participants) | 17 | 9
score
  Baseline (n=16,8) | 53.71 (19.881) | 59.24 (15.350)
  Day 85 (n=17,8) | 14.51 (22.319) | 53.53 (29.817)

ADVERSE EVENTS:
Time Frame: 1 year 5 mos
Groups:
- IGE025 300mg: IGE025 administered subcutaneously every 4 weeks at the study center
- Placebo: Placebo administered subcutaneously every 4 weeks at the study center.
Arm/Group | IGE025 300mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/10
Other Adverse Events (participants affected / at risk) | 17/20 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGE025 300mg (N=20) | Placebo (N=10)
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IGE025 300mg (N=20) | Placebo (N=10)
Constipation (Gastrointestinal disorders) | 1 | 0
Tongue pruritus (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 7 | 3
Periodontitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0
Fungal test positive (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1
Haematoma (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.